CLINICAL TRIAL: NCT00925340
Title: Effects of the Family Check-Up on Adolescents With Alcohol-Related Events and Their Siblings
Brief Title: Family Check-Up for Adolescents and Siblings
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Brown University (Other)
Collaborators: National Institute on Alcohol Abuse and Alcoholism (NIAAA) (NIH)
Responsible Party: Principal Investigator, Anthony Spirito, Professor, Brown University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NIAAA-Spirito-AA017659; R01AA017659 (NIH); NIH Grant 1R01 AA017659-01
Record Dates: First submitted 2009-06-19; First posted 2009-06-22 (Estimated); Last update posted 2014-07-29 (Estimated); Status verified 2014-07

CONDITIONS: Alcohol Abuse
Keywords: Alcohol; Substance Abuse; Adolescent; Family functioning
MeSH Terms: conditions — Alcoholism; Substance-Related Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 - Family Check Up (Experimental): Brief family intervention that employs Motivational Interviewing.
  Interventions: Behavioral: Family Check Up
- 2 - Psychoeducation (Active Comparator)
  Interventions: Behavioral: Psychoeducation

INTERVENTIONS:
Behavioral: Family Check Up — The Family Check-Up provides a thorough assessment of individual family strengths and weaknesses and utilizes principles of motivational interviewing to encourage families to change.
  Arms: 1 - Family Check Up
Behavioral: Psychoeducation — Psychoeducation regarding teen alcohol and drug use in general, along with ways parents can help their children stay safe from using alcohol or drugs.
  Arms: 2 - Psychoeducation

SUMMARY:
A two group randomized design will be used to test the primary hypothesis that the experimental intervention will reduce alcohol consumption and alcohol-related negative consequences significantly more than a comparison family-based psychoeducation condition in both an identified alcohol-using adolescent (12- 18 years old) and his/her teenage sibling (the sibling can be 3 years older or younger than teen with the sibling's age between 12-21 years old). The experimental condition consists of the Family Check-up, while the comparison condition is a less intense parenting psychoeducation program. Time points will include follow-ups at 3, 6, and 12 months.

DETAILED DESCRIPTION:
A total of 175 adolescents, 12 to 18 years old, will be drawn from multiple sites to compare the experimental condition, The Family Check Up(FCU; Dishion & Kavanagh, 2003) to a family-based psychoeducational program.

The Family Check-Up is a selective intervention program that focuses on parents. Its goal is to provide individualized feedback to motivate parents to make improvements in their parenting practices. A unique strength of the FCU is that feedback is individualized and tailored to specific parenting skills as they typically pertain to an identified adolescent in the family. We propose to evaluate the efficacy of the FCU when applied to both an adolescent identified patient (IP) and a sibling close in age. Our rationale for including a sibling close in age derives from a strong empirical base which has shown that: 1) sibling resemblance for alcohol use is high and environmental factors shared by siblings account for substantial portions of variance in adolescent alcohol use; and 2) specific interactional dynamics of the sibling relationship (collusion) are related to teen alcohol use. Dr. Dishion has found that in high-risk families, sibling collusion accounts for variance in problem behavior after controlling for involvement with deviant peers. This connection between ineffective parenting strategies and sibling relationship dynamics in combination creates increased risk for alcohol use by siblings close in age. This notion serves as a foundation to examine the efficacy of a sibling-enhanced FCU intervention with respect to: 1) improvement in parental communication and monitoring; 2) reduction of sibling interactive behaviors that are associated with alcohol use; and 3) reduction of alcohol use in IP adolescents as well as siblings who are currently using alcohol. We will test specified mediators of FCU efficacy in reducing levels of alcohol use at both the parenting level and at the level of sibling dynamics. In order to determine whether other types of family-based interventions might be just as helpful as the more intensive FCU, efficacy of the sibling-enhanced FCU will be compared to a parenting psychoeducational program.

ELIGIBILITY:
Inclusion Criteria:

* Participants will be 12 to 18 years old, inclusive, living at home with at least one parent or guardian.
* Participants will have a teenage sibling within 3 years of age of the identified adolescent patient. Siblings can be either biological or unrelated siblings in blended families, as long as they live in the same home as the parents targeted in the intervention conditions. The adolescent must have experienced a recent (within 1 month) alcohol-related event (ED admission, school disciplinary action, grounding by parents, legal action). The adolescent must also screen in by reaching the clinical cutoff score on the Adolescent Drinking Index.

Exclusion Criteria:

* Alcohol positive adolescents with substance dependence diagnosis requiring a higher level of care; 18 year olds living on their own.

Ages: 12 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 104 (Actual)
Dates: Start 2008-09; Primary Completion 2014-07 (Actual); Study Completion 2014-07 (Actual)

PRIMARY OUTCOMES:
Teen and sibling alcohol use | 3 months
  drinking frequency (days per month), quantity (drinks per occasion), frequency of high-volume drinking (5 or more drinks per occasion)
Teen and sibling alcohol use | 6 months
  drinking frequency (days per month), quantity (drinks per occasion), frequency of high-volume drinking (5 or more drinks per occasion
Teen and sibling alcohol use | 12 months
  drinking frequency (days per month), quantity (drinks per occasion), frequency of high-volume drinking (5 or more drinks per occasion

SECONDARY OUTCOMES:
Teen and sibling marijuana use | 3 months
  Days of marijuana use in prior 3 months
Teen and sibling marijuana use | 6 months
  Days of use in prior 3 months
Teen and siblings marijuana use | 12 months
  Days of use in prior 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Anthony Spirito, PhD, Principal Investigator — Brown University
Locations (1):
- Brown University, Providence, Rhode Island, United States

REFERENCES:
- [Derived] Spirito A, Hernandez L, Marceau K, Cancilliere MK, Barnett NP, Graves HR, Rodriguez AM, Knopik VS. Effects of a brief, parent-focused intervention for substance using adolescents and their sibling. J Subst Abuse Treat. 2017 Jun;77:156-165. doi: 10.1016/j.jsat.2017.02.002. Epub 2017 Mar 2. PMID 28259500